CLINICAL TRIAL: NCT00054743
Title: Global Initiative to Characterize Differences in Antiretroviral Pharmacokinetics in HIV-Infected Populations
Brief Title: Differences in Blood Levels of Nevirapine in HIV-infected Patients in Uganda and the United States
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030091; 03-CC-0091
Record Dates: First submitted 2003-02-07; First posted 2003-02-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-28

CONDITIONS: HIV Infection
Keywords: Race; Ethnicity; Pharmacogenetics; Cytochrome P450; Population Pharmacokinetics; HIV
MeSH Terms: conditions — HIV Infections | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood draw

SUMMARY:
This study will determine whether blood levels of the anti-HIV medicine nevirapine are different in HIV-infected patients in the United States from patients in Uganda. People from all over the world take medications to treat HIV infection. These medicines work well in some people but not in others, and they cause harmful side effects in some people and not in others. These differences may be related to variations in how much of the drug reaches the blood. Differences in drug blood levels among people in various areas of the world may be attributed to differences in diet, state of health, ability to absorb the medicines from the stomach, ability to eliminate the drugs from the body, and the brand of medicine taken. This study will help scientists learn whether differences in blood levels of HIV medicines are important in determining how well the drugs work in different patient populations.

HIV-infected patients 18 years of age and older in the United States and in Kampala, Uganda who have been on an antiretroviral treatment regimen that includes at least 28 consecutive days of nevirapine may be eligible for this study. Candidates will be screened with a medical history, physical examination, and blood tests.

Participants will have a total of approximately about 5 ounces of blood drawn during this 6- to 8-hour study. They will come to the NIH clinic in the morning, and a catheter (plastic tube) will be inserted into an arm vein for collecting blood. (Alternatively, blood can be collected by a needle inserted into an arm vein.) Blood will be withdrawn according to the following schedule:

* About 5 tablespoons will be collected upon arrival at the clinic after an overnight fast. Within 30 minutes of this blood draw, the patient will have breakfast and take his or her morning dose of nevirapine, along with any other medications that need to be taken at that time.
* 1 tablespoon of blood will be drawn 2 hours after the nevirapine dose.
* 1 tablespoon of blood will be drawn 4 hours later (6 hours after the nevirapine dose).

The blood will be analyzed for levels of nevirapine and possibly other HIV medicines. Some of the blood will be stored for later analysis of genes (cytochrome P450 and MDR1) that are involved in eliminating medicines from the body.

...

DETAILED DESCRIPTION:
The overwhelming majority of HIV-infected persons reside in the developing world. As such, recent efforts have focused on providing antiretroviral pharmacotherapy to this population. However, there are a number of factors indigenous to non-Western HIV-infected patients that may alter their virologic, immunologic, and/or toxicologic response to antiretroviral therapy. Absorption, distribution, and clearance of antiretroviral medications may differ among patients residing in non-Western countries secondary to dietary influences, parasitic infection, and malabsorption. Genetic polymorphisms of drug metabolizing enzymes (cytochrome P450; CYP) and drug transporters (i.e. P-glycoprotein) may also contribute to altered pharmacokinetics among these patients. The purpose of this pilot, hypothesis-generating study is (1) to characterize the pharmacokinetics of the non-nucleoside reverse transcriptase inhibitor nevirapine in a non-Western HIV-infected population (Kampala, Uganda) and in a similar cohort of HIV-infected individuals in the United States and (2) to compare pharmacokinetic parameter values between the groups. Twenty-five subjects from each site will participate. Subjects from the Ugandan site may participate regardless of their CD4+ lymphocyte count and viral load; they will be studied prior to the U.S. cohort. The U.S. group will be selected to include subjects that are matched by gender to their Ugandan counterparts. Subjects will have one pre-dose and two post-dose blood samples collected for the determination of nevirapine plasma concentrations. Samples will be analyzed using LC/MS-MS. Population pharmacokinetics parameter values (Cmax, Cmin, AUC, CL/F, Vd) will be determined using NONMEM(Trademark) and compared between groups. Blood samples collected during the study will also be used to determine CYP and MDR1 genotypes of study subjects in an effort to explain any observed differences in pharmacokinetics parameter values between the study populations.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Documentation in the patient's medical record of HIV-1 infection using double ELISA or a second confirmatory test (e.g., Western Blot) or any one of the following: detectable p24 antigen, quantifiable plasma HIV RNA, or detectable proviral DNA.
  2. Males and females greater than or equal to 18 years of age
  3. Laboratory values within acceptable limits

     AST/SGOT less than or equal to 5 times the upper limit of normal (ULN)

     Serum creatinine less than or equal to 2 times the ULN

     Hemoglobin greater than or equal to 9.0 g/dL
  4. Receipt of a stable nevirapine-containing antiretroviral regimen for at least 28 days.
  5. Informed consent signed and subject declares that they have been adherent to their nevirapine-containing antiretroviral regimen.

EXCLUSION CRITERIA:

1. Presence of life-threatening or unstable renal, hepatic, cardiovascular, hematologic, neurologic, psychiatric, or respiratory disease, as determined by medical records, or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigator.
2. Laboratory values outside acceptable limits

   AST/SGOT less than 5 times the upper limit of normal (ULN)

   Serum creatinine greater than 2 times the ULN

   Hemoglobin less than 9.0 g/dL
3. Positive pregnancy test.
4. Receipt of IL-2 within 3 months of study participation.
5. Drug or alcohol use that may impair safety or adherence.
6. Poor venous access.
7. Documented or reported fever (greater than 38.5 degrees C) within 7 days of screening.
8. Active opportunistic infection requiring therapy.
9. Refusal to agree to allow for specimens to be stored for future research.
10. Greater than 4 loose/soft stools per day.
11. Subject is non-adherent with their nevirapine-containing antiretroviral regimen and/or they have not provided informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-02-06; Study Completion 2011-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Joint Clinical Research Center (JCRC), Kampala, Uganda

REFERENCES:
- [Background] Danner SA, Carr A, Leonard JM, Lehman LM, Gudiol F, Gonzales J, Raventos A, Rubio R, Bouza E, Pintado V, et al. A short-term study of the safety, pharmacokinetics, and efficacy of ritonavir, an inhibitor of HIV-1 protease. European-Australian Collaborative Ritonavir Study Group. N Engl J Med. 1995 Dec 7;333(23):1528-33. doi: 10.1056/NEJM199512073332303. PMID 7477167
- [Background] Harris M, Durakovic C, Rae S, Raboud J, Fransen S, Shillington A, Conway B, Montaner JS. A pilot study of nevirapine, indinavir, and lamivudine among patients with advanced human immunodeficiency virus disease who have had failure of combination nucleoside therapy. J Infect Dis. 1998 Jun;177(6):1514-20. doi: 10.1086/515317. PMID 9607828
- [Background] Hoetelmans RM, Reijers MH, Weverling GJ, ten Kate RW, Wit FW, Mulder JW, Weigel HM, Frissen PH, Roos M, Jurriaans S, Schuitemaker H, de Wolf F, Beijnen JH, Lange JM. The effect of plasma drug concentrations on HIV-1 clearance rate during quadruple drug therapy. AIDS. 1998 Jul 30;12(11):F111-5. doi: 10.1097/00002030-199811000-00002. PMID 9708400